CLINICAL TRIAL: NCT02832284
Title: Feasibility Study of a Bronchoscopic Ultrasound-Guided Tissue Acquisition System With Real-time Visualization for Collection of Cytology Specimens of Peripheral Pulmonary Lesions
Brief Title: iNod System Human Feasibility Assessment
Acronym: iNod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E7113
Record Dates: First submitted 2016-06-27; First posted 2016-07-14 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Solitary Pulmonary Nodule; Biopsy, Fine-Needle
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- iNod System (Experimental): Multi-center, Prospective, Single-arm Feasibility Study with Salvage.
  Interventions: Device: iNod System

INTERVENTIONS:
Device: iNod System — The iNod System is intended for use for diagnostic ultrasound imaging and ultrasound-guided fine needle aspiration (FNA) of extramural and submucosal lesions of the tracheobronchial tree.

SUMMARY:
The purpose of this study is to demonstrate feasibility to access, visualize, and obtain specimens adequate for cytology of lung lesions in subjects with suspected lung cancer when using the iNod System.

DETAILED DESCRIPTION:
This protocol is a traditional feasibility study for the sampling of a peripheral pulmonary lesion in the setting of a suspicion of lung cancer. Standard of practice radial endobronchial ultrasound (R-EBUS) transbronchial needle aspiration (TBNA) is visualizing a peripheral lesion on R-EBUS, locking the placement of the access sheath, removing the ultrasound catheter from the access sheath and then blindly advancing a sampling device to acquire cellular matter for cytologic evaluation. The iNod system performs the same procedure with one fewer device exchange. It provides real-time visualization of the biopsy needle and target peripheral pulmonary lesions during tissue acquisition. The ultrasound probe is not retracted in advance of the sampling maneuver and the sampling is completed under direct visualization. Compared to current standard of care methods for transbronchial sampling of pulmonary lesions, this approach is not expected to add additional risk. Tissue sampling under real-time visualization may improve the efficiency of tissue sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 18 years or older.
2. Subject is willing and able to comply with study procedures and provide written informed consent to participate in study.
3. Subject with a predominantly solid lung lesion, 1 cm to 7 cm in diameter, which has been identified on chest CT (obtained within 6 weeks) with the intention to undergo a clinically indicated bronchoscopic evaluation under routine clinical care. If the lesion is partially solid (i.e. there is a ground glass component) then the solid portion must make up 80% of the lesion.
4. Subject for whom the decision to pursue biopsy has been made by the treating physician and agreed upon by the subject.

Exclusion Criteria:

1. Subjects with pure ground glass opacity, a subsolid target lesion, and/or a ground glass opacity identified on Chest CT.
2. Subjects with lesions that include endobronchial involvement, per Chest CT.
3. Subjects who lack fitness to undergo flexible bronchoscopy and standard of care Radial EBUS-guided cytological assessment evaluations, as determined by the investigator.
4. Subjects with known coagulopathy.
5. Subjects who are pregnant or nursing mothers.
6. Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bowman, MD, Study Director — Medical Director, Boston Scientific
Locations (3):
- United States (3):
  - Johns Hopkins University Medical School, Baltimore, Maryland
  - Washington University of St. Louis, St Louis, Missouri
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-policy.html).
Supporting Information: Study Protocol, SAP
Time Frame: The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-policy.html).
Access Criteria: The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-policy.html).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iNod System
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 23 Patients were analyzed for primary endpoint. 86 Attempts to access target lesions were analyzed.
Units Other Than Participants: Attepmts at target lesions
Groups:
- iNod System: Multi-center, Prospective, Single-arm Feasibility Study with Salvage.
  iNod System: The iNod System is intended for use for diagnostic ultrasound imaging and ultrasound-guided fine needle aspiration (FNA) of extramural and submucosal lesions of the tracheobronchial tree.
  Per, protocol, each of the 23 enrolled subjects underwent evaluations with the iNod System.
  For study subjects for whom an adequate specimen, defined as a specimen that has been confirmed as suitable for cytologic evaluation, is not obtained from the iNod System diagnostic procedure but for whom continuation with endobronchial maneuvers are not contraindicated, additional standard of care (SOC) R-EBUS-guided diagnostic sampling maneuvers should be conducted.
Arm/Group | iNod System
Number analyzed (Participants) | 23
Number analyzed (Attepmts at target lesions) | 86
Age, Continuous [Mean (Full Range); unit: years] | 68.0 [48.0 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Acquisition of Adequate Specimens of Targeted Lung Lesions
Description: The primary endpoint for the iNod Feasibility Study was clinical success, defined as the iNod System's ability to acquire adequate specimens of cellular matter suitable for the cytologic evaluation of targeted lung lesions, under real-time visualization.
Time Frame: Intraprocedural
Measure: Count of Participants; unit: Participants
Arm/Group | iNod System
Number analyzed (Participants) | 23
Participants | 9

2. Secondary Outcome: Device/Procedure-Related Safety Events
Description: Occurrence and severity of Adverse Events related to the iNod System biopsy procedures, as well as Adverse Events related to any subsequent Radial EBUS-guided salvage procedures.
Time Frame: Procedure through Post-procedure call; 6-8 days post-procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | iNod System
Number analyzed (Participants) | 23
Participants | 6

3. Secondary Outcome: Visualization
Description: Lesions visualized during iNod Maneuvers
Time Frame: Intraprocedural
Population: Lesions visualized per attempt to visualize lesion
Measure: Count of Units; unit: Lesions visualization attempts
Units Other Than Participants: Lesions visualization attempts
Arm/Group | iNod System
Number analyzed (Participants) | 23
Number analyzed (Lesions visualization attempts) | 86
Lesions visualization attempts | 72

4. Secondary Outcome: Access
Description: Lesions accessed where iNod Biopsy Needles were deployed in the target lesion during study maneuvers
Time Frame: Intraprocedural
Population: Lesions accessed per attempt to access lesion
Measure: Count of Units; unit: Lesions access attempts
Units Other Than Participants: Lesions access attempts
Arm/Group | iNod System
Number analyzed (Participants) | 23
Number analyzed (Lesions access attempts) | 86
Lesions access attempts | 72

5. Secondary Outcome: Acquisition
Description: iNod maneuvers that acquired specimens of cellular matter for cytology
Time Frame: Intraprocedural
Population: Specimens of cellular matter for cytology per attempt, to acquire cellular matter.
Measure: Count of Units; unit: Specimens of cellular matter for cytolog
Units Other Than Participants: Specimens of cellular matter for cytolog
Arm/Group | iNod System
Number analyzed (Participants) | 23
Number analyzed (Specimens of cellular matter for cytolog) | 78
Specimens of cellular matter for cytolog | 69

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the Baseline/Consenting Visit, through study exit; typically 7 days.
Description: Any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons, whether or not related to the investigational medical device.
  NOTE 1: This includes events related to the investigational medical device or comparator.
  NOTE 2: This definition includes events related to the procedures involved (any procedure in the clinical investigation plan).
Arm/Group | iNod System
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iNod System (N=23)
Pseudomonas Pneumonia (Infections and infestations) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iNod System (N=23)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was not powered or designed as a study of diag. yield. Nor was this study designed to follow pts. with indeterminate cytology diagnoses. Non-malig. cytopathology. findings would require 6 mos. of follow-up (min. expect.) for a yield study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT02832284/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT02832284/SAP_001.pdf